CLINICAL TRIAL: NCT01978847
Title: Proposal for Retrospective Review of Anterior&Posterior Cervical, Thoracic, and Lumbar Instrumented Arthrodesis Surgeries Performed at OSU.
Brief Title: Retrospective Review of Anterior and Posterior Cervical, Thoracic, and Lumbar Instrumented Arthrodesis Surgeries
Status: Completed | Type: Observational
Sponsor: H Francis Farhadi, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, H Francis Farhadi, MD, PhD, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2013H0153
Record Dates: First submitted 2013-10-24; First posted 2013-11-08 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Spinal Condition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective review will allow for an evaluation of potential patient- or procedure-related factors that are associated with the development of either radiologic or clinical adjacent-segment pathology.

DETAILED DESCRIPTION:
Spinal arthrodesis can be performed through either anterior, posterior, or lateral approaches for a variety of traumatic, degenerative, or deformity conditions. In recent years, the development of more sophisticated segmental instrumentation techniques and hardware has allowed for incorporation of multiple spinal levels in single settings. The long-term consequences for spinal motion segments adjacent to such fusions remain unknown.

The investigators propose to undertake a retrospective case study analysis evaluating both radiologic and clinical parameters indicative of adjacent-segment pathology in patients who have undergone instrumented arthrodesis procedures at Ohio State University, performed by either Dr. Francis Farhadi, James B. Elder, or Gary Rea.

ELIGIBILITY:
Inclusion Criteria:

* Must have had a Spinal arthrodesis procedure at Ohio State University

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal arthrodesis can be performed through either anterior, posterior, or lateral approaches for a variety of traumatic, degenerative, or deformity conditions.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-05; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
The number of patients with radiologic evidence of fusion | 5 years
  Radiologic review will include X-Rays, CT, and MRI at pre-surgery, as well as X-rays at 6 weeks, 3, 6, 12, 24, 36, 48 and 60 months post-operatively.

SECONDARY OUTCOMES:
The number of patient with clinical evidences of fusions | 5 years
  examples of clinical measurement are Pain Scores and the Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Francis Farhadi, MDPHD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Unviersity, Columbus, Ohio, United States